CLINICAL TRIAL: NCT00708357
Title: Does eNOS Gene Polymorphism Play a Role in the Maintenance of Basal Vascular Tone in the Choroid or Optic Nerve Head?
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc Prof Priv.-Doz. Dr, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: OPHT-311004
Record Dates: First submitted 2008-06-26; First posted 2008-07-02 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Ocular Physiology; Regional Blood Flow
Keywords: eNOS Gene Polymorphism; ocular blood flow
MeSH Terms: interventions — omega-N-Methylarginine

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Other): homozygous mutant: CC allele of the eNOS T-786C gene
  Interventions: Drug: NG-monomethyl-L-arginine
- 2 (Other): homozygous mutant: TT allele of the eNOS T-786C gene
  Interventions: Drug: NG-monomethyl-L-arginine

INTERVENTIONS:
Drug: NG-monomethyl-L-arginine — intravenous administration, bolus over 5 minutes, dosage 6mg/kg
  Other Names: L-NMMA

SUMMARY:
Nitric oxide (NO) is a potent endothelium-derived vasodilatator that plays a major role in the control of ocular blood flow. Endothelial NO synthase (eNOS) is one of three isoforms of NOS producing NO through hydroxylation of L-arginine. The eNOS gene is located on the long arm of chromosome 7, and different polymorphic variations have been identified. These single nucleotide polymorphisms (sNP´s) have the ability to change transcription activity and therefore enzyme levels. Recent data indicate that the T -786C polymorphism (especially the homozygous variant) is associated with reduced eNOS activity and consequently impaired NO production.

In the present study the investigators want to investigate if the T -786C eNOS gene polymorphism determines choroidal and optic nerve head blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Homozygous variants of the T -786C genotyping (CC or TT)
* Normal ophthalmic findings, ametropia less than 3 diopters

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-05; Primary Completion 2009-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Genotyping | performed during the first year before measurements

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Department of CLinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria